CLINICAL TRIAL: NCT06786299
Title: Clinical Study on the Safety and Efficacy of Autologous CD84 Chimeric Antigen Receptor T-Cell Therapy for Adult Relapsed/Refractory Acute Myeloid Leukemia.
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: BRL Medicine Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: [2024]TXB NO.019
Record Dates: First submitted 2025-01-02; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Relapsed/Refractory Acute Myeloid Leukemia(AML)
Keywords: Relapsed/Refractory Acute Myeloid Leukemia(AML); CD84 Chimeric Antigen Receptor T-Cell Therapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD84-CART therapy arm (Experimental)
  Interventions: Biological: RD-IIT-001; Drug: CD84-CART

INTERVENTIONS:
Biological: RD-IIT-001 — Autologous CD84 Chimeric Antigen Receptor T-Cell Therapy
Drug: CD84-CART — Autologous CD84 Chimeric Antigen Receptor T-Cell Therapy

SUMMARY:
Acute Myeloid Leukemia (AML) is an aggressive type of leukemia, with high relapse rate and poor long term survival in adults. Traditional treatment regimens mainly include chemotherapy and hematopoietic stem cell transplantation. In the past decade, with the application of molecular targeted drugs and immunotherapy, the survival of AML patients has significantly improved. Relapsed/refractory (R/R)-AML is a state following the failure of AML treatment, with more complex therapy and poorer prognosis, necessitating more clinical trials and new treatment methods to improve patients' survival and quality of life. In this study, we propose a treatment approach that include therapying with autologous CD84 chimeric antigen receptor T-cell. Our study aims to answer the safety and efficacy of this treatment regimen, and further improve the survival for those participants.

DETAILED DESCRIPTION:
This is a non-randomized, open-label, single-arm clinical study. A total of 12-18 adults aged 18-70 with relapsed/refractory acute myeloid leukemia (AML) participants will be enrolled. The primary endpoint is maximal tolerable dose(MTD), recommended phase II dose, and dose limiting toxicity (28 Days).

The research process includes the screening period, apheresis period, lymphocyte depletion preconditioning period, treatment observation period, and follow-up period.

Screening period (from signing the informed consent form to D-29):

After the subject signs the informed consent form and before the apheresis period, various tests are conducted according to the requirements of the screening period. Subjects who fully meet the inclusion criteria and do not meet the exclusion criteria at all are included in the study.

Apheresis period (D-28):

After signing the informed consent form, eligible subjects need to undergo peripheral blood mononuclear cell (PBMC) collection before treatment, using a component blood collection method to circulate and collect no less than 1×10^9 cells of PBMC to prepare RD-IIT-001.

Lymphocyte depletion preconditioning period (D-5 to D-1):

Five days before the first infusion of RD-IIT-001, a preconditioning assessment is conducted. After the assessment, qualified subjects undergo lymphocyte depletion preconditioning treatment before the first infusion of RD-IIT-001. The lymphocyte depletion preconditioning regimen is as follows:

Fludarabine: 25 mg/m2, Day(D)-5, D-4, D-3, for three consecutive days by intravenous infusion; Cyclophosphamide: 300 mg/m2, D-5, D-4, for two consecutive days by intravenous infusion.

Or the dosage of the lymphocyte depletion regimen may be adjusted according to the absolute value of peripheral blood lymphocytes.

After lymphocyte depletion preconditioning, an assessment is conducted on D-1 before the infusion of RD-IIT-001. For subjects who are not suitable for the infusion of RD-IIT-001, the infusion may be suspended, and the infusion may be postponed for up to 7 days after the end of the lymphocyte depletion treatment.

Treatment observation period (D0 to D28):

After completing the assessment before the infusion of RD-IIT-001, qualified subjects receive a single one-time intravenous infusion of RD-IIT-001 on D0. Subjects who receive RD-IIT-001 infusion need to be observed in the hospital for at least 14 days. Those with a suitable donor and deemed eligible for transplantation by the study will proceed to undergo allogeneic hematopoietic stem cell transplantation. If not transplanted, patients will be followed up on D21 and D28 for safety and efficacy-related examinations. The period from the day of RD-IIT-001 infusion to day 28 (±3 days) is the DLT observation period.

Follow-up period (D29 to M24):

Starting from the second month after the first infusion of RD-IIT-001 and ending at the 24th month, the follow-up period involves assessing the effectiveness and safety of the subjects as well as survival follow-up according to the trial process schedule.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-70 years (inclusive of boundary values), gender unrestricted.
2. Voluntarily participate in this clinical study, sign the informed consent form, have good compliance, and cooperate with follow-up visits.
3. Diagnosed with relapsed/refractory acute myeloid leukemia (AML), patients with relapsed/refractory AML must meet one of the following conditions: patients who have not achieved remission after two standard treatment courses; relapse within 12 months after complete remission; relapse after 12 months but have not achieved remission after one standard treatment; patients with second or subsequent relapses. Relapse is defined as the reappearance of leukemia cells in the peripheral blood or the presence of ≥5% blasts in the bone marrow (excluding other causes such as bone marrow regeneration after consolidation chemotherapy) or the infiltration of leukemia cells in extramedullary sites after achieving complete remission (CR) of AML, excluding cases where the above conditions occur after granulocyte colony-stimulating Factor （G-CSF） treatment.
4. Flow cytometry confirms the presence of CD84-positive blasts.
5. ECOG (Eastern Cooperative Oncology Group) score of 0-1.
6. Able to collect T cells that meet the required specifications.
7. Liver Function: Alanine Aminotransferase (ALT) ≤ 3 × Upper Limit of Normal (ULN); Aspartate Aminotransferase (AST) ≤ 3 × ULN; Total Bilirubin (TBIL) ≤ 1.5 × ULN (except in cases of Gilbert's syndrome).
8. Renal Function: Creatinine Clearance Rate (CrCl) ≥ 60 ml/minute (Cockcroft/Gault formula).
9. Coagulation Function: International Normalized Ratio (INR) ≤ 1.5 × Upper Limit of Normal (ULN), Prothrombin Time (PT) ≤ 1.5 × ULN.
10. Cardiac Function: Hemodynamic stability is good, with a Left Ventricular Ejection Fraction (LVEF) ≥ 50%.
11. Pulmonary Function: No clinically significant pleural effusion, baseline oxygen saturation >92%.
12. Female subjects of childbearing potential and male subjects with partners of childbearing potential must use medically recognized contraceptive measures or abstain from sexual activity during the study treatment period and for at least 6 months after the study treatment ends. Female subjects of childbearing potential must have a negative serum human chorionic gonadotropin （HCG） test within 7 days prior to study enrollment and must not be breastfeeding.

Exclusion Criteria:

1. Individuals with a history of severe drug allergies or allergic constitution;
2. Those with uncontrolled active infections;
3. Individuals with severe cardiac diseases, such as angina, myocardial infarction, heart failure, and arrhythmias;
4. Subjects with congenital immunoglobulin deficiencies;
5. Patients with other malignant tumors (except for non-melanoma skin cancer, carcinoma in situ of the cervix, bladder cancer, and breast cancer with more than 5 years of disease-free survival);
6. Subjects with end-stage renal failure;
7. Subjects who are positive for Hepatitis B surface antigen (HBsAg) or Hepatitis B core antibody (HBcAb) with peripheral blood HBV DNA levels above the detection limit; those positive for Hepatitis C virus (HCV) antibody with peripheral blood HCV RNA positivity; individuals positive for Human Immunodeficiency Virus (HIV) antibody; and those with positive syphilis tests;
8. Individuals with mental illnesses and severe cognitive impairments;
9. Those who have participated in other clinical trials within the last month;
10. Pregnant or breastfeeding women;
11. Subjects deemed inappropriate for the study by the investigator or for other reasons not suitable for inclusion in this study;
12. Recipients of allogeneic transplants who relapsed within three months or still have graft-versus-host disease (GVHD) reactions more than three months after the transplant;
13. Central nervous system leukemia involvement.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-02-10 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximal tolerable dose (MTD）; Recommended phase II dose (RP2D）; Dose limiting toxicity （DLT） | 28 days ±3 days
  Dose limiting toxicity (DLT) is defined as an adverse event that is judged to be definitely or possibly related to RD-IIT-001, occurring from the first infusion of RD-IIT-001 up to Day 28 (±3 days). Safety evaluations are conducted using the NCI-CTCAE 5.0 criteria.
  Maximal tolerable dose (MTD）：Three dose levels （1.0×10^6 cells/kg；3.0×10^6 cells/kg；6.0×10^6 cells/kg）are preset, with the observation period for dose-limiting toxicity (DLT) from the first infusion of RD-IIT-001 up to Day 28 (±3 days). Dose escalation follows the "3+3" design principle.
  Recommended phase II dose (RP2D）：After completing dose escalation, 3-6 additional subjects may be enrolled at the MTD dose level to determine the RP2D. If the MTD dose level has not been reached, the investigator may decide, based on PK and efficacy data, whether to increase to a higher dose or expand with 3-6 3-6 additional subjects at the current highest dose level to determine the RP2D.

CONTACTS AND LOCATIONS:
Locations (1):
- No. 79, Qingchun Road, Hangzhou City, Zhejiang Province., Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided